CLINICAL TRIAL: NCT05931328
Title: A Single-arm, Prospective, Multicenter Clinical Trial of the Combination of Thiotepa and Pomalidomide for the Treatment of Relapsed/Refractory Primary Central Nervous System Lymphoma.
Brief Title: The Study of the Combination of Thiotepa and Pomalidomide for the Treatment of Relapsed/Refractory Primary Central Nervous System Lymphoma Patients.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJ-RR-PCNSL-01
Record Dates: First submitted 2023-06-27; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Relapsed or Refractory (R/R) Primary Central Nervous System Lymphoma
MeSH Terms: conditions — Recurrence | interventions — pomalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- thiotepa+pomalidomide (Experimental): thiotepa combined with pomalidomide: thiotepa 30mg/m2,intravenously guttae, on day 1; pomalidomide 12mg orally daily for 2 weeks. A chemotherapy cycle lasts for 3 weeks.
  Interventions: Drug: thiotepa combined with pomalidomide

INTERVENTIONS:
Drug: thiotepa combined with pomalidomide — thiotepa combined with pomalidomide: thiotepa 30mg/m2,intravenously guttae, on day 1; pomalidomide 12mg orally daily for 2 weeks. A chemotherapy cycle lasts for 3 weeks.

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of the combination of thiotepa and pomalidomide in the treatment of relapsed/refractory (R/R) primary central nervous system lymphoma (PCNSL).

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed PCNSL, diagnosed according to the 2016 WHO diagnostic criteria. Previously treated with at least one course of chemotherapy, with disease progression or recurrence.

Aged 18 to 75 years old; ECOG PS score of 0 to 4 points; Expected survival time of more than 3 months; A whole-body PET/CT and head MR (plain scan + enhancement) performed within 28 days before study enrollment should show at least one measurable lesion in two perpendicular directions (based on the 2014 Lugano criteria), or abnormal findings in cerebrospinal fluid examination (including cerebrospinal fluid cells, NGS), or ocular examination confirming lesions in the retina or vitreous body;

Adequate organ function, defined as follows:

Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Renal function: serum creatinine (Cr) ≤ 1 × ULN or creatinine clearance rate (CCR) ≥ 90 mL/min; Cardiac function: cardiac function grade of III or less (NYHA standard); echocardiography shows an ejection fraction of ≥50%; Coagulation function: international normalized ratio (INR) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 10s, and prothrombin time (PT) ≤ 3s; Thyroid function: baseline thyroid-stimulating hormone (TSH) level is normal or baseline TSH is abnormal, but T3/T4 is normal and there are no symptoms; Women of childbearing age must take contraceptive measures or undergo a pregnancy test with a negative result before enrollment, and take contraceptive measures during the trial and within 90 days after the last dose of the drug; for men, contraceptive measures must be taken during the trial and within 90 days after the last dose of the drug, or they must have undergone surgical sterilization; The subject voluntarily agrees to participate in the study, signs an informed consent form, has good compliance, and cooperates with follow-up.

Exclusion Criteria:

Pregnant or lactating women; Patients with involvement of sites other than the central nervous system; Patients with bone marrow failure, specifically defined as absolute neutrophil count (ANC) <1.5 x 109/L, platelets <75 x 109/L, and hemoglobin <70 g/L;

Patients diagnosed with malignant tumors other than lymphoma or currently undergoing treatment, with the following exceptions:

* Patients who have received curative treatment and have not had any known active malignant tumors for ≥5 years prior to enrollment; ② Patients with adequately treated basal cell carcinoma of the skin without evidence of disease (excluding melanoma); ③ Patients with adequately treated cervical intraepithelial neoplasia without evidence of disease.

Known allergy to any component of the investigational drug; Patients who have undergone allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; Patients who may receive other systemic anti-tumor therapy during the study period; Patients with human immunodeficiency virus (HIV) antibodies, active hepatitis, or other uncontrolled infectious diseases; Patients with a history of clear neurological or psychiatric disorders; Patients who may interfere with the participation of the subject in the study or the evaluation of study results due to drug abuse, medical, psychological or social conditions; Patients deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to 2 years.
  The proportion of subjects who achieves a best overall response of CR or PR.
Adverse event rate | Baseline up to 3 years.
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).

SECONDARY OUTCOMES:
2-year Progression-free Survival (PFS) rate | Baseline up to 2 years.
  The proportion of patients who did not experience disease progression at 2 years.
2-year Overall Survival（OS）rate | Baseline up to 3 years.
  The proportion of patients who survived at 2 years.
Duration of Response（DOR） | Baseline up to 2 years.
  From the date that CR or PR are first occurred to the date of objective disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province People's Hospital., Nanjing, Jiangsu, China